CLINICAL TRIAL: NCT00776672
Title: The Objective of This Study is to Compare the Relative Bioavailability of Fosinopril Sodium 40 mg Tablets (Ranbaxy Laboratories Limited, Lot No. 1238312) With That of Monopril® in Healthy Adult Subjects Under Non-Fasting Conditions
Brief Title: Bioequivalence Study of Fosinopril 40mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy research laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B025508
Record Dates: First submitted 2008-10-17; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Fosinopril Tablets
MeSH Terms: interventions — Fosinopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): fosinopril sodium 40 mg tablets of Ranbaxy
  Interventions: Drug: Fosinopril 40mg Tablets
- 2 (Active Comparator): Monopril® 40mg tablets
  Interventions: Drug: Fosinopril 40mg Tablets

INTERVENTIONS:
Drug: Fosinopril 40mg Tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of fosinopril sodium 40 mg tablets (Ranbaxy Laboratories Limited, Lot No. 1238312) with that of Monopril® in healthy adult subjects under non-fasting conditions.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomised, two-treatment, two-period, two-sequence, single-dose, crossover , bioequivalence study on Fosinopril formulations comparing fosinopril 40mg tablets of Ranbaxy Laboratories with Monopril®, in healthy, adult, human, subjects under non-fasting conditions

Eligible subjects underwent pre-study examinations that included a physical examination, 12-lead ECG, and laboratory tests - including hematology, blood chemistries, urinalysis, infectious diseases (Hepatitis B, Hepatitis C, HIV), and urine drUgs of abuse. Laboratory testing for female subjects also included a serum pregnancy test.

Twenty four (24) subjects were enrolled in this study; 23 completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized subjects consisting of members of the community at large.

Characterization of Study Group

* All subjects selected for this study will be at least 18 years of age.
* Clinical laboratory measurements will include the following:

Hematology:

* hemoglobin, hematocrit,
* red blood cell count,
* platelets, and white blood cell count (with differential).

Clinical Chemistry:

* creatinine, BUN, glucose, SGOT/AST,
* SGPT/ALT, bilimbin, and alkaline phosphatase.

Urine Analysis:

* pH, specific gravity, protein, glucose,
* ketones, bilimbin, occult blood, and cells.

HIV Screen:

* (pre-study only) Hepatitis-B, C Screen:
* (pre-study only) Drugs of Abuse Screen: pre-study and at check-in each study period

Exclusion Criteria:

* Subjects with a history of chronic alcohol consumption (during past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma(during past 5 years),diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested (including any penicillin product) should be excluded from the study.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at check-in each study period. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drag within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (eg condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives (except Lunelle monthly injection) anytime during the 6 months prior to study dosing, Lunelle monthly injection anytime during the 45-days prior to study dosing or used hormonal contraceptives within 14 days before dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check in in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-10; Primary Completion 2002-10 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html